CLINICAL TRIAL: NCT05202587
Title: The Evaluation of the Agreement and Precision of the Notal Vision Home OCT in the Automatic Fluid Quantification in Patients With NV-AMD.
Brief Title: The Evaluation of the Agreement Between the NVHO in the Automatic Fluid Quantification and Cirrus OCT
Status: Completed | Type: Observational
Sponsor: Notal Vision Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C2021.006
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Neovascular Age-related Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multi-center study will enroll Adult subjects diagnosed with neo-vascular age-related macular degeneration (NV-AMD) in at least one eye at the time of enrollment. the subject study duration for this study is one day (2-3 hours). Each study site will have two NVHO devices and one Cirrus 5000 and the patients will be scand on the two NVHO devices and one Cirrus device as a part of the study flow. At the Study Visit, fluid must be present in approximately 280 study eyes and fluid must be absent from 20 study eyes. Each subject will only have one study eye. The fluid status will be determined by the investigator while reviewing an acceptable screening Cirrus OCT volume scan.

DETAILED DESCRIPTION:
Screening will include refraction, best corrected visual acuity and Cirrus OCT. Subjects will receive a general overview of the self-operation of the NVHO system. The general overview will include written material and a verbal explanation.

If only one eye qualifies for enrollment, that eye will be assigned as the study eye. If both eyes are eligible, the study eye will be assigned according to a randomization schedule unless the fluid type (IRF or SRF) between eyes is different, in which case the randomization can be overridden at the discretion of an Investigator to fulfill the required sample size of the fluid type. volume scans will be calculated for each enrolled eligible study eye Once the study eye has been identified, the subject will be assigned to either perform a Cirrus OCT first or perform self-imaging on a NVHO first. The order between the Cirrus OCT or the NVHO will be assigned according to a randomization schedule. Whichever is assigned first will be completed followed by the second assigned device.

Cirrus OCT Scans:

When the study eye is assigned to perform the Cirrus OCT, the study eye will be scanned, non-dilated with a Cirrus 5000 OCT device, up to 4 times with the objective of obtaining two acceptable volume scans for the study eye. The enrolled subjects that are randomized to have Cirrus volume scans first will be discontinued before NVHO self-imaging if two acceptable Cirrus volume scans cannot be obtained.

NVHO Scans:

When the study eye is assigned to perform the NVHO OCT scans, the subject will:

1. Be escorted to a separate room, with two NVHO devices.
2. Be given an explanation of the procedure of self-imaging 4 repeated NVHO volume scans from each of the two NVHO devices. The order of the two NVHO devices will be assigned according to a randomization schedule.
3. Perform a tutorial on the better seeing eye as indicated by the subject on the first randomly assigned device, even if this better seeing eye is not the study eye.
4. Perform a successful calibration on the study eye in up to 3 attempts on the first NVHO device. In case of 3 repeated failures in calibration, the participation of the subject in the study will be terminated.
5. Self-image the study eye 4 times on the first NVHO device (in order to have at least 3 images eligible for NOA fluid quantification), with a short break between scans.
6. When 4 images are obtained on the first device, perform a successful calibration on the second NVHO device with the study eye in up to 3 attempts. In case of 3 repeated failures in calibration, the participation of the subject in the study will be terminated.
7. Self-image the study eye 4 times on the second NVHO device, with a short break between scans.
8. When 4 scans are obtained on both NVHO devices, scanning is completed.

Subject Exit from the Study:

After the subject has completed all the study procedures, the subject will be discontinued from the study. Subjects may withdraw voluntarily from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ability to speak, read and understand English. 2. Ability to understand and agree to contents of informed consent either in writing or verbally.

  3. Adult diagnosed with NV-AMD in at least one eye with or without fluid based on the subject's medical record.

  4. Best corrected Visual Acuity of 20/320 or better in the study eye. 5. Available and willing to conduct Cirrus imaging and NVHO self-imaging in a clinic environment.

Note: Eyes with other pathologies including pseudocysts, outer retinal tubulations, pigment epithelial detachments, hemorrhage, subretinal hyper-reflective material (SHRM), geographic atrophy, sub-retinal pigment epithelium (RPE) hypo-reflective areas, epiretinal membrane (ERM), macular hole, and hyperreflective retinal spots (Foci) can be enrolled.

Exclusion Criteria:

* 1. Any other retinal disease requiring steroid or anti-VEGF injections. 2. Cirrus scan during screening with Signal Strength <6. 3. Dry AMD in study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll approximately 140 AMD patients diagnosed with NV-AMD presenting with IRF and 140 AMD patients presenting with SRF in at least one eye at the time of enrollment, and 20 eyes with no fluid for a total of 300 subjects
Sampling Method: Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Intra-Retinal Fluid (IRF) | 5 minutes
  volume [nl] of the Intra-retinal fluid
Sub-Retinal Fluid (SRF) | 5 minutes
  volume [nl] of the Sub-retinal fluid
IRF spatial distribution | 5 minutes
  frontal view (en-face) of IRF thickness map
SRF spatial distribution | 5 minutes
  frontal view (en-face) of SRF thickness map
IRF area segmentation | 5 minutes
  Segmented B-scans of the IRF
SRF area segmentation | 5 minutes
  Segmented B-scans of the ISRF
Mean central retinal thickness | 5 minutes
  Retina thickness (µ) in 5 central ETDRS grid fields (Total, superior, temporal, inferior, nasal, and central)

CONTACTS AND LOCATIONS:
Overall Officials: Gidi Benyamini, Study Director — Notal vision Druyanov 5, Tel Aviv
Locations (5):
- United States (5):
  - Brian Joondeph, Lakewood, Colorado
  - Florida Retina Institute, PA, Orlando, Florida
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Tennessee Retina, PC, Nashville, Tennessee
  - Strategic Clinical Research Group, Willow Park, Texas

IPD SHARING:
Plan to Share IPD: Undecided